CLINICAL TRIAL: NCT05673733
Title: Additional Effects of Scapular Stabilization Exercise With Exergaming Training on Upper Limb Functions in Chronic Stroke Patients
Brief Title: Additional Effects of Scapular Stabilization Exercise With Exergaming Training in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Shumailakiran
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Exergaming Training
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Exergaming training combined with Scapular stabilization exercises will be performed for 6 weeks for 3 times per week.
  Interventions: Other: scapular stabilization exercises with exergaming training
- Group B (Active Comparator): Exergaming training will be performed for 6 weeks for 3 times per week.
  Interventions: Other: exergaming training

INTERVENTIONS:
Other: scapular stabilization exercises with exergaming training — Group A will receive scapular stabilization exercises with exergaming training
  Arms: Group A
Other: exergaming training — Group B will receive only exergaming training
  Arms: Group B

SUMMARY:
The World Health Organization has termed stroke to be a clinical syndrome, of presumed vascular origin, typified by rapidly developing signs of focal or global disturbance of cerebral functions and the leading cause of death worldwide in 2016 making it a major non-contagious cause of death. This study would be beneficial in a way that it will give a valuable input and will contribute for the knowledge of interventions for stroke with an emphasis on upper extremity function among health care practitioners for their goal of promoting health, prevention of diseases and improving quality of life.

DETAILED DESCRIPTION:
Exergaming can contribute to improvement of the function of UE motor and AROM in chronic stroke patients, additional studies with a large number of subjects with long follow-up periods are required to determine their effectiveness neurorehabilitation stimulation . The exergaming protocol presented in this study represents success a tool for UE functional aspects in patients with chronic stroke. It has shown improvement in gripping strength, handicrafts and UE's operational recovery. Movement control and the position of scapula determine an optimal upper limb function. Paresis leading to scapular disorientation ultimately exaggerates motor impairment in upper extremities. Recent literature has emphasized on the need to design an upper extremity protocol including scapular stabilization exercises in order to increase muscular strength and decrease scapular dyskinesis .The results of a study showed that scapular stability exercises had an impact on hand function and the ability to move hemiplegic patients after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stroke patients with an initial onset of 6 months or above.
* Those who had 30-65 points by Fugl-Meyer Assessment of upper extremity
* Those who had minimum score 24 on mini mental state examination
* Those who have the ability to execute at least 20' of active shoulder flexion and abduction against gravity those who could understand and follow instructions provided by the investigator
* Those who are medically stable enough to participate in active rehab
* Those who have no problems with auditory or visual functioning.
* Modified Ashworth Scale (MAS) 1-3

Exclusion Criteria:

* Orthopaedic or mental health problems
* Those who have difficulty to stay in a sitting position
* Severe conditions such as uncontrolled blood pressure or angina
* History of epilepsy
* The refusal to play a video game.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment tool of Upper Extremity Function | 2 months
  To assess motor functioning, balance , sensation and joint functioning in patients with post-stroke hemiplegia.
  Change from baseline and 2 months
Wolf Motor Function Test | 2 months
  It quantifies upper extremity (UE) motor ability through timed and functional tasks. The items are rated on a 6-point scale.
  Change from baseline and 2 months
Jebsen Taylor Hand Function Test | 2 months
  It is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).
  - Scoring: The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, stimulated feeding, stacking, and lifting large, lightweight, and heavy objects. Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.
  Change from baseline and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Shumaila, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No